CLINICAL TRIAL: NCT06874478
Title: The Rate and Predictors of Respiratory Distress Among Neonates Delivered by Elective Cesarean Section at Term
Brief Title: Respiratory Distress and Elective Cesarean Section at Term
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Professor, Assiut University
Other Study IDs: RD-CS
Record Dates: First submitted 2025-03-08; First posted 2025-03-13 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with gestational age ≥ 37 weeks who will be delivered by elective cesarean section: Those women will be subjected to pulmonary artery doppler velocimetery
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — The main pulmonary artery will be seen between the pulmonary valve and the bifurcation of the right and left branches. The pulsed Doppler sample gate will be adjusted to 3 mm, and the angle of insonation will be kept at or around 15°. Doppler gain and scale will be tailored for optimizing the velocity waveform display, clearly showing the peak systolic velocity (PSV) and early diastolic notch. The MPA Doppler waveform will show a sharp systolic peak blood flow with a needle-like appearance. After the optimum fetal main pulmonary artery waveform, Doppler velocity will be manually traced three times, and the average will be taken.

SUMMARY:
Cesarean section is a life-saving surgical operation for women and their newborns. In Egypt, caesarean sections are over-utilized. The rate increased from 27.6 % in 2008 to 51.8 % in 2014, reaching 72.2 % in 2021. Cesarean section has been associated with an increased risk of adverse respiratory outcomes in newborns. Studies have shown a higher risk of neonatal respiratory distress syndrome in babies born by elective cesarean section, especially at 37 and 38 weeks' gestation. Neonatal respiratory distress syndrome is one of the leading causes of neonatal morbidity and mortality. Many non-invasive tools have been used to predict the risk of neonatal respiratory distress syndrome. Most of these studies assessed the predictors of neonatal respiratory distress syndrome in low birth or preterm fetuses, and none of them talked about neonatal respiratory distress syndrome with term fetuses. Doppler velocimetry provides a simple and non-invasive method to assess the fetal pulmonary circulation. Pulmonary Doppler velocimetry is used to determine lung maturity in complicated pregnancies. The magnitude of neonatal respiratory distress syndrome among term neonates depends on the availability of medical services and the number of trained medical personnel. So, there is a need to assess the rate and predictors of eonatal respiratory distress syndrome among low-risk term fetuses delivered by Cesarean section to give attention and appropriate intervention for these predictors to decrease the morbidity and mortality associated with eonatal respiratory distress syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Maternal age of 20-39 years.
2. Women with singleton pregnancy ≥ 37 weeks
3. Pregnant women who received corticosteroid to enhance lung maturity and will be subjected to elective cesarian section (before onset of labour) within 1 week after administration of corticosteroid

Exclusion Criteria:

1. Women with oligohydramnios or polyhydramnios.
2. Women with underlying disease requiring corticosteroids.
3. Pregnant women with any medical disorders such as hypertension, diabetes, renal diseases, antiphospholipid syndrome, intrauterine growth restriction, preterm premature rupture of membrane, placenta previa, antepartum haemorrhage, on anticoagulant thereby.
4. Women with confirmed fetal malformation.
5. Women who will refuse to participate.

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Woman who will be delivered by cesarian section at term
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
the rate of neonatal respiratory distress syndrome by pulmonary artery velocimetry | 37 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Woman's Health Hospital - Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes